CLINICAL TRIAL: NCT07315932
Title: Current Knowledge and Perceptions of Hormone Replacement Therapy Among Patients Aged 11 to 18 Years, and Their Parents, Treated for Hypogonadism at the Strasbourg University Hospital
Brief Title: Perception of Hormonal Replacement Therapy Among Patients Aged 11 to 17 Years
Acronym: THS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9620
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Female Hypogonadism
Keywords: Female Hypogonadism; Central hypogonadism; Peripheral hypogonadism; hormone replacement therapy
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish a current knowledge and perception of patients and their parents regarding HRT in order to assess the needs that can promote understanding and adherence to treatment by implementing therapeutic education workshops

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 11 to 18 years
* Treated at the University Hospital of Strasbourg for central or peripheral hypogonadism with the initiation of hormone replacement therapy

Exclusion Criteria:

- Inability to provide the subject with clear information (difficulties understanding the subject, language barrier, illiteracy, etc.)

Ages: 11 Years to 18 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Female patients aged 11 to 18 years treated at the University Hospital of Strasbourg for central or peripheral hypogonadism with the initiation of hormone replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of patients' knowledge about the composition of hormonal treatment for female hypogonadism | Up to 7 months
  The aim is to assess the knowledge of patients aged 11 to 18 about the composition of hormone treatment for female hypogonadism using a questionnaire.
Assessment of patients' knowledge regarding the effects of hormonal treatment for female hypogonadism | Up to 7 months
  The aim is to assess the knowledge of patients aged 11 to 18 years about the effects of hormone treatment for female hypogonadism using a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie et obstétrique - CHU de Strasbourg - France, Strasbourg, France